CLINICAL TRIAL: NCT01428141
Title: A Phase I Study of E7050 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7050-J081-110
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Solid Tumor; Gastric Cancer
Keywords: Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms; Gastrointestinal Neoplasms | interventions — N-(2-fluoro-4-((2-(4-(4-methylpiperazin-1-yl)piperidin-1-yl)carbonylaminopyridin-4-yl)oxy)phenyl)-N'-(4-fluorophenyl)cyclopropane-1,1-dicarboxamide

ARMS (1):
- E7050 (Experimental)
  Interventions: Drug: E7050

INTERVENTIONS:
Drug: E7050 — Drug: E7050 The starting dose of E7050 will be 400 mg given orally, once-daily, in patients with advanced tumor that have progressed following effective therapy. The study consists of 2 parts: a Tolerability Confirmation Component to confirm the tolerable dose in subjects with solid tumor and an Expansion Component to confirm the safety and to preliminarily assess the anti-tumor activity in subjects with gastric cancer.

SUMMARY:
The purpose of this study is to investigate the tolerability, safety, pharmacokinetics (PK), pharmacodynamics (PD) and anti-tumor activity of E7050 when administered orally once daily to patients with advanced solid tumor and gastric cancer.

ELIGIBILITY:
Inclusion Criteria

1. Aged from 20 to less than 75 years old at the time of obtaining informed consent.
2. Histological or cytological diagnosis of solid tumors.
3. Subjects who have progressed after treatment with approved therapies or for whom there are no standard effective therapies available.
4. Adequate organ function.
5. Subjects who have no carryover of effect from prior therapy or no adverse drug reactions (excluding alopecia) that may affect the safety evaluation of the investigational drug.
6. Performance Status (PS) 0-1 established by Eastern Cooperative Oncology Group (ECOG).
7. Expected to survive for 3 months or longer after starting administration of the investigational drug.

Exclusion Criteria

1. Females who are pregnant or breastfeeding.
2. Brain metastases with clinical symptoms or which requires treatment.
3. Serious complications or disease history.
4. Subjects who cannot take oral medication.
5. Using antiplatelet/anticoagulant drugs.
6. Continuous using of drugs or foods that strongly inhibit or induce CYP3A4/5 or CYP2D6 during the study period.
7. Scheduled for surgery during the study period.
8. Known to be HIV, HBV or HCV positive.
9. Suffering from psychotic disorder(s) and/or unstable recurrent affective disorder(s) evident by use of anti-psychotics or have had a suicide attempt(s) within approximately the last 2 years.
10. History of drug or alcohol dependency or abuse within 2 years.
11. Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
12. Received any other investigational product or device within 4 weeks before administration.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose (MTD) | During the Run-in Phase and Cycle 1 period (the first 5 weeks of treatment)
  Determination of the MTD of E7050 given orally once daily. MTD is the highest dose at which no more than 1 out of 6 patients experiences dose-limiting toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Obaishi, Study Director — Japan/Asia Clinical Research Product Creation Unit, Eisai Co., Ltd.
Locations (3):
- Japan (3):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Sunto, Shizuoka